CLINICAL TRIAL: NCT02193698
Title: Single Arm Open-label Trial to Investigate the Efficacy and Safety of Lenlidomide as a Treatment for Recurrent or Refractory Crow-Fukase (POEMS) Syndrome
Brief Title: Efficacy and Safety of Lenalidomide as a Treatment for Recurrent or Refractory POEMS Syndrome Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Sonoko Misawa, Associate Professor, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G26007
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: POEMS Syndrome
Keywords: POEMS syndrome; lenalidomide
MeSH Terms: conditions — POEMS Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide+Dexamethasone (Experimental): Cycle1 : Lenalidomide 15mg/day (day 1-21) Cycle2-6 : Lenalidomide 25mg/day (day 1-21) Dexamethasone 20mg/day (day 2. 9, 16, 23)
  Interventions: Drug: Lenalidomide+Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide+Dexamethasone — Lenalidomide 25mg/day (day 1-21) Dexamethasone 20mg/day (day 2. 9, 16, 23)
  Other Names: Lebramide+Decadoron

SUMMARY:
This study investigates the efficacy and safety of Lenalidomide as a treatment for recurrent or refractory POEMS (Crow-Fukase) syndrome.

DETAILED DESCRIPTION:
This study investigates the efficacy and safety of Lenalidomide as a treatment for recurrent /refractory POEMS (Crow-Fukase) syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Crow-Fukase syndrome (confirmed by diagnostic criteria.)
2. Recurrent or refractory Crow-Fukase syndrome.
3. Patients without severe liver or renal dysfunction.
4. Patients without severe neutropenia or thrombocytopenia.
5. Patients without clinically problematic ECG findings
6. Negative on the pregnacy test on the day 1 of cycle 1.
7. Patients who can undertake prevention of pregnancy, if necessary.
8. Patients with written informed consent.
9. Patients who are capable of ambulatory hospital visits every 4 weeks.
10. Patients with informed consent to the registration and rules of RevMate®.

Exclusion Criteria:

1. Patients who have been administered, bortezomib, lenalidomide, melpharan within 4 weeks prior to the registration.
2. Patients who have been on steroid treatment (more than 10mg/day in predonine) within 2 weeks prior to the registration.
3. Patients who have been administered bevacizumab within 12 weeks prior to the registration.
4. Patients who could worsen acutely during the clinical trial period.
5. Patients with severe complicaitons ( cardiac failure, renal failure liver failure, bleeding enterogastric ulcer, ileus, poorly controlled diabetes.
6. Patients with malignancies.
7. Female patients who are pregnant or desire childbearing. Males who desire fertility.
8. Patients who allergic to lenalidomide or dexamethasone.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reduction rate of serum VEGF | after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonoko Misawa, MD, Principal Investigator — Chiba University, Department of Neurology
Locations (1):
- Chiba University Graduate School of Medicine Department of neurology, Chiba, Chiba, Japan